CLINICAL TRIAL: NCT03263845
Title: Round-trip Survey or Urine Bag: Evaluation of Pain in Urinary Collections in Pediatric Emergencies in Children Who Have Not Acquired Cleanliness (SONDAPU)
Brief Title: Evaluation of Pain in Urinary Collections in Pediatric Emergencies in Children Who Have Not Acquired Cleanliness
Acronym: SONDAPU
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3036_SONDAPU
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Urinary Tract Infections in Children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study.

DETAILED DESCRIPTION:
Febrile urinary infections account for 5% of unexplained causes of fever in children up to 2 years of age. Urinary samples are therefore very common in pediatric emergencies. In children who have not acquired cleanliness, the most used method of collection is the placement of a sterile urine bag on the perineum. It allows a noninvasive urinary collection. However from a bacteriological point of view this method is debatable because the rate of contamination of the collections is important. This mode of collection is of interest only to exclude a urinary infection, by the realization of a urinary strip.

Pocket-collected urine is not reliable for bacteriological analysis in culture. For example, if the urine strip is positive, the American Academy of Pediatrics recommends urine sampling by urine sampling (or other invasive methods) for culture.

The urine bag should be changed every 30 minutes to avoid the risk of contamination. The technique is wait-and-see, the installation of several pockets is often necessary before obtaining urine.

A study carried out in 2014 shows that in 39.4% of the cases the withdrawal of the urinary pouch was as much more painful than the urinary sounding, in the same patient. To our knowledge there is no other study dealing with the difference in pain engendered by these two methods.

Since the urinary catheterization is faster, bacteriologically justified and necessary if the pocket collection is positive, it seems legitimate to ask ourselves if we should not aim at a generalization of the urinary catheterization, as first intention, Having not acquired cleanliness, requiring a withdrawal of urine for suspicion of urinary infection.

Many centers continue to use urinary pocket collection mainly, as the survey technique seems too invasive and painful.

ELIGIBILITY:
Inclusion Criteria:

Children under 3 years of age who have not acquired the cleanliness present at the pediatric emergency department in Rennes, where urine sampling is necessary in case of suspected urinary tract infection.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under 3 years of age who have not acquired the cleanliness present at the pediatric emergency department in Rennes, where urine sampling is necessary in case of suspected urinary tract infection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain | Day 0
  Score of the visual analog scale rated by the caregiver during the first performed gesture.

SECONDARY OUTCOMES:
Evaluation of pain | Day 0
  Score of the visual analog scale rated by the parent during the first performed gesture.
Evaluation of pain | Day 0
  Score of the visual analog scale rated by the parent and the caregiver for the following gestures
The experience of the gesture by the parent and the caregiver | Day 0
  Evaluation by a questionnaire by choosing from the following proposals:
  Very well spent, well spent, badly spent or very badly spent
Time needed to collect urine | Day 0
  Duration between the first gesture and the final urine collection

CONTACTS AND LOCATIONS:
Overall Officials: Amelie Rickewaert, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France